CLINICAL TRIAL: NCT06914401
Title: Oxygenation Procedure for Obese Patients Using High Flow Oxygen Therapy Combined With Non-invasive Ventilation During Intubation in the Operating Room: a Randomised Controlled Trial
Brief Title: Oxygenation Procedure for Obese Patients During Intubation in the Operating Room
Acronym: POP-OVNI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A02304-43
Record Dates: First submitted 2025-03-28; First posted 2025-04-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia Induction
Keywords: Non Invasive Ventilation; High Flow Nasal Oxygen; Intubation; Obese
MeSH Terms: conditions — Obesity | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined oxygenation procedure (Active Comparator)
  Interventions: Procedure: NIV (Non Invasive Ventilation) and HFNO (High Flow Nasal Oxygen)
- Single oxygenation procedure (Active Comparator)
  Interventions: Procedure: NIV (Non Invasive Ventilation)

INTERVENTIONS:
Procedure: NIV (Non Invasive Ventilation) and HFNO (High Flow Nasal Oxygen) — Combination of two procedures Preoxygenation prior to intubation with NIV (Non Invasive Ventilation) and HFNO (High Flow Nasal Oxygen).
  During intubation, NIV is stopped and apneic oxygenation is maintained with HFNO
  Arms: Combined oxygenation procedure
Procedure: NIV (Non Invasive Ventilation) — Single procedure Preoxygenation prior to intubation with NIV (Non Invasive Ventilation).
  Arms: Single oxygenation procedure

SUMMARY:
Obesity is a risk factor for difficult intubation, with an incidence of up to 15.5%, and difficult mask ventilation. Obesity also reduces the functional residual capacity (FRC) of the lungs, the main reservoir of oxygen during apnoea. Complications associated with induction and intubation in the operating room are more frequent in obese patients. Preoxygenation is a cornerstone in the management of patients at risk of desaturation during induction. The study aims to compare two oxygenation strategies , in obese patients. Oxygenation using a combination of NIV (Non Invasive Ventilation) and HFNO (High Flow Nasal Oxygen) compared with NIV alone in the operating room for induction of general anaesthesia with orotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring general anaesthesia with orotracheal intubation in the operating room
* Obese patient (Body Mass Index , BMI ≥ 30kg/m2)
* Patient affiliated to or benefiting from a social security scheme
* Patient having signed the free and informed consent form.

Exclusion Criteria:

* Haemodynamic instability
* Intubation without laryngoscopy (fibroscope intubation) or nasotracheal intubation
* Emergency surgery not allowing patient consent.
* Patient with a contraindication to NIV or OHD
* Protected patients: Adults under guardianship, curatorship or other legal protection; deprived of liberty by judicial or administrative decision; pregnant, breast-feeding or parturient women; hospitalised without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Oxygen reserve | 2 minutes after intubation
  The lowest level of end-tidal oxygen concentration (EtO2)

SECONDARY OUTCOMES:
SpO2 | during preoxygenation; before intubation; during intubation; after intubation; 2 minutes after intubation
  Peripheral oxygen saturation
Rate of EtCO2 | 2 minutes after intubation
  End-tidal carbon dioxide
Patient tolerance | Day 2, at study end
  Numerical Rating Scale (NRS)
  [minimum value 0, maximum value 10] higher score mean a better outcome
Adverse events | Perioperative/Periprocedural
  moderate and severe complications

CONTACTS AND LOCATIONS:
Overall Officials: Ségolène MROZEK, MD, PhD, Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France

IPD SHARING:
Plan to Share IPD: No